CLINICAL TRIAL: NCT01436292
Title: Hypoalbuminemia in Burn Patients: Should we Care? - A Randomized Controlled Clinical Pilot Trial
Brief Title: Hypoalbuminemia in Burn Patients
Acronym: Halburns
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No funding
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE 10.239
Record Dates: First submitted 2011-07-14; First posted 2011-09-19 (Estimated); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Second or Third Degree Burns
Keywords: Hypoalbuminemia; Burns; Albumin; Organ dysfunction; Outcome
MeSH Terms: conditions — Neoplasm Metastasis; Hypoalbuminemia; Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Albumin (Experimental): Patient will receive 5% HAS daily for the first 7 days of stay in ICU according to their albumin level
  Interventions: Drug: 5% human albumin solution (HAS)

INTERVENTIONS:
Drug: 5% human albumin solution (HAS) — Patient will receive 5% HAS daily for the first 7 days of stay in ICU according to their albumin level:
  ≥ 30 gr/L: albumin will not be administered; 25 - 29.9 gr/L: 25 g of 5% HAS; 20 - 24.9 gr/L: 50 g 5% HAS; 15 - 19.9 gr/L: 75 g of 5% HAS; 10 - 14.9 gr/L: 100 g of 5% HAS; < 10 gr/L: 150 g of 5% HAS.

SUMMARY:
The purpose of this study is to determine whether 5% human albumin solution, given to correct hypoalbuminemia, could improve organ dysfunction in burn patients as assessed by a change in the SOFA score from baseline to day 7 (or before if the patient is discharged from the ICU or died).

DETAILED DESCRIPTION:
Each year approximately 2 million people are burned in the USA, from which 80,000 are hospitalized and 6,500 die. It is a well known fact that the two most important factors for mortality in burn patients are age and percent total body surface area burn (TBSA), which are unmodifiable findings.

A predictable inflammatory response takes place after a burn injury leading to profound changes in patient homeostasis. As a result, hypoalbuminemia is one of the common finding in severe burn patients. 21% of hospitalized adult patients are hypoalbuminemic on admission. After admission, worsening of existing hypoalbuminemia and development of de novo one are frequently seen.

Moreover, hypoalbuminemia, a potentially modifiable variable, has been strongly associated with poor clinical outcomes in critically ill patients and in burn patients.

Dynamic organ dysfunction scores have been introduced in critically ill patients few years ago in order to describe the evolution of patients on a daily basis. The Sequential Organ Failure Assessment (SOFA) score is now one of the most accepted score in critically ill patients and has been validated in general medico-surgical unit, as well as in trauma and cardiac surgery patients. It encompasses components assessing six organ functions. This score has also been shown to predict mortality in critically ill patients and in burn patients when used in a dynamic way.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to the BICU in the Centre hospitalier de l'Université de Montréal within 24 hours following their thermal burn injury.
2. Patients with second or third degree burns greater or equal than 20% of total body surface area.
3. Patients aged 18 years or older. -

Exclusion Criteria:

1. Patients with serum albumin greater than 30 g/dl at the time of randomization.
2. Patients with a do not resuscitate order.
3. Patients needing total parenteral nutrition.
4. Patients with the following chronic diseases that could affect baseline SOFA calculation or serum albumin levels: end-stage kidney disease, nephrotic syndrome, hepatitis, exudative enteropaty, chronic thrombocytopenia or hematological malignancy.
5. Patients with a known reaction to albumin.
6. Pregnant or lactating women.
7. Patients younger than 18 years old. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Organ dysfunction as assessed by a change in the SOFA score from baseline to day 7 (or before if the patient is discharged from the ICU or died). | Seven days

SECONDARY OUTCOMES:
ICU and hospital mortality | 1, 3 and 6 months
ICU and hospital length of stay | 1, 3 and 6 months
Free days of mechanical ventilation | Seven days
Caloric intake | Seven days
Fluid balance | Seven days
Incidence of infection | Seven days
Time to complete coverage defined as the time between admission and last surgery for grafting | 1, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Eljaiek, MD, Principal Investigator — Université de Montréal - CHUM; Marc-Jacques Dubois, MD - FRCPC, Principal Investigator — Université de Montréal - CHUM
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada